CLINICAL TRIAL: NCT02763943
Title: Improving Medication Safety and Cardiovascular Risk Factor Control in Kidney Transplant Recipients
Brief Title: Improving Medication Safety and CVD Risk Factor Control in Kidney Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Prevention
Other Study IDs: Pro00051804
Record Dates: First submitted 2016-03-14; First posted 2016-05-05 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2016-04

CONDITIONS: Cardiovascular Diseases; Diabetes Mellitus; Medication Adherence
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Medication Adherence

INTERVENTIONS:
Behavioral: Pharmacist-led, technology enabled education intervention — Prospective, non-randomized, pilot study assessing the feasibility and potential efficacy of a 6-month, pharmacist-led, technology enabled education intervention on improving medication safety and cardiovascular risk factor control in adult solitary kidney transplant recipients with a secondary aim of assessing if the impact of the intervention varies by race.

SUMMARY:
There is a lack of data analyzing the influence of Cardio-vascular Diseases (CVD) risk factor control on graft survival disparities in Black transplant recipients. Studies in the general population indicate that CVD risk factor control is poor in Black patients, leading to higher rates of renal failure and CV events. However, with the exception of hypertension, there is paucity in data demonstrating similar results within transplant recipients. Recent analyses conducted within our transplant program, indicate that CVD risk factors, especially diabetes, are poorly controlled in Black recipients, which likely impacts graft loss. Since these data were collected in a retrospective manner, larger analyses are needed to validate these exploratory findings.

This pilot study is to:

1. Determine if the study is feasible, as measured by the proportions of enrolled to approached and completed to enrolled.
2. Measure and compare, at baseline versus the end of the intervention, the medication safety events, including the number of medication errors, medication non-adherence and medication side effects, in patients enrolled in the study
3. Measure and compare, at baseline versus the end of the intervention, CVD risk factor control, including hypertension, diabetes and dyslipidemia, in patients enrolled in the study
4. Measure and compare, at baseline versus the end of the intervention, patient reported survey results, in patients enrolled in the study
5. Determine if the impact of the intervention is more pronounced in Black recipients, as compared to non-Black recipients

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age and able to give informed consent.
2. Received a first or repeat cadaveric or living donor renal transplant.
3. Patient has adequate graft function, defined as an estimated glomerular filtration rate (GFR) of at least 20 mL/min, using the 4-variable Modification of Diet in Renal Disease (MDRD) equation.
4. Patient is at least one year post transplant.
5. Patient has documented hypertension, defined as a sitting blood pressure of at least 140/90 mmHg or receiving any anti-hypertensive therapy.
6. Patient has documented diabetes mellitus, defined as a hemoglobin A1c of at least 6.5% or receiving any anti-glycemic medications.
7. Willing to comply with all study visits.

Exclusion Criteria:

1. Biopsy proven acute rejection episode that occurred within the past month.
2. Patients who have received an organ transplant other than a kidney.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-01-22 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure values from baseline to end of study | 6 months
  Blood pressure will be assessed using clinic measurements, taken three times, five minutes apart in the same arm and averaged.
Change in HBA1C values from baseline to end of study | 6 months
Change in lipid values from baseline to end of study | 6 months
Medication adherence by comparing medication possession ratios (MPR) for the six months prior to enrollment compared to six months during the intervention | 1 year
Patient self-reported medication adherence at baseline compared to end of study. | 6 months
  The Morisky 8-item adherence score will be compared from baseline to end of study.
Number of medication errors assessed at baseline and compared to errors at 6 months | 6 months
Medication side effects at baseline compared to end of study. | 6 months
  The Memphis side effect scale will be used to compare side effects from baseline to end of study.
Patient reported survey results regarding self-care and health knowledge from baseline to end of study | 6 months
Patient reported survey results regarding psychosocial status from baseline to end of study | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Taber DJ, Gebregziabher M, Posadas A, Schaffner C, Egede LE, Baliga PK. Pharmacist-Led, Technology-Assisted Study to Improve Medication Safety, Cardiovascular Risk Factor Control, and Racial Disparities in Kidney Transplant Recipients. J Am Coll Clin Pharm. 2018 Dec;1(2):81-88. doi: 10.1002/jac5.1024. Epub 2018 Jun 21. PMID 30714026